CLINICAL TRIAL: NCT00362830
Title: A Study of the Alternating Administration of Ixabepilone and Vinflunine Every Three Weeks in Patients With Advanced Cancer
Brief Title: A Study of the Alternative Administration of Ixabepilone and Vinflunine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA183-008
Record Dates: First submitted 2006-08-07; First posted 2006-08-10 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — vinflunine; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: vinflunine + ixabepilone

INTERVENTIONS:
Drug: vinflunine + ixabepilone — solution for injection, IV, vinflunine: 250 to 320 mg/m2 + ixabepilone: 30 to 40 mg/m2, every 3 wks, variable duration

SUMMARY:
The purpose of the study is to test how vinflunine interacts with ixabepilone in the human body.

ELIGIBILITY:
Inclusion Criteria:

* ECOG status of 0-1

Exclusion Criteria:

* Inability to tolerate venous access
* Brain mets
* Severe nerve damage
* ANC <2,000/mm3
* Platelets <100K
* Bilirubin >= 1.5 times the IULN
* ALT/AST >= 2.5 times the IULN
* Creatinine <50 mL/min
* Prior treatment with vinflunine and/or ixabepilone
* Strong use of CYPP450 drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and describe any dose limiting toxicities of ixabepilone and vinflunine in an alternating regimen. | upon occurrence

SECONDARY OUTCOMES:
Determine the overall safety profile, efficacy and rate and extent to which ixabepilone and vinflunine are absorbed or otherwise available to the treatment site in the body. | upon occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - University Of Miami Miller School Of Medicine, Miami, Florida
  - The Cleveland Clinic Foundation, Cleveland, Ohio